CLINICAL TRIAL: NCT01134783
Title: Evaluating Innovative Weight Reduction Strategies for College Students
Brief Title: Choosing Healthy Options in College Environments and Settings
Acronym: CHOICES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 0908S71521; 1U01HL096767 (NIH)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): The CHOICES intervention included a 1-credit, academic college course focusing on healthy weight behaviors and participation in a social networking and social support website
  Interventions: Behavioral: CHOICES Intervention
- Control Group (No Intervention): Control group (serving as a comparison group)

INTERVENTIONS:
Behavioral: CHOICES Intervention — Academic course on healthy weight behaviors followed by participation in a social networking and social support website.
  Arms: Intervention Group

SUMMARY:
Examine the effectiveness of a weight gain prevention intervention to positively affect body mass index in 2-year college students

DETAILED DESCRIPTION:
The goal of this research is to develop and test innovative strategies to help prevent unhealthy weight gain in college students attending 2-year community or technical colleges. The intervention we propose for Phase 2, and will refine through our formative experiences in Phase 1, will be based on social ecological and social networks models with students randomized to conditions. Students (n=440) with BMIs between 20.0 and 34.9 will be recruited to participate in an intervention trial that lasts 24 months. After the initial screening and consent procedures, students will complete baseline measures that include: assessment of body composition; blood pressure and a blood draw; a behavioral and psychosocial survey; medical and weight history and two 24-hour online dietary recalls. After the completion of baseline assessments, students will be randomized into treatment or control conditions. Students randomized into the intervention condition will participate in a 1-credit course offered through their 2-year college that focuses on eating, activity, sleep and stress management as ways to help maintain or achieve a healthy weight; three course sections will be offered to accommodate students' scheduling needs and learning preferences. A web-based social network and support component will be introduced as part of this course and will continue as the intervention channel for 20 months following the 1-credit course. This supported intervention phase will use a study-designed website to reinforce, inform and encourage exchange and support between all intervention participants. Students will be asked to track their weight and weight-control behaviors on the website and intervention staff will interact with participants electronically or through phone calls offering encouragement and helping with problem solving. Control students will receive their health assessments and usual care including existing public health information on maintaining a healthy weight and information regarding health services offered on their school's campus. The effectiveness and sustainability of the intervention approaches will be evaluated.

The primary aim is to examine the effectiveness of a 24-month weight gain prevention intervention to positively affect BMI in 2-year college students. Our hypothesis is that students randomized to an intervention condition will experience a smaller increase in mean BMI post treatment, as compared to students randomized to the control condition.

The secondary aims of this study are to: 1) Examine the effectiveness of a weight gain prevention intervention to positively affect weight in 2-year college students' and 2) compare the effects of the intervention and control groups with regard to change in BMI and weight from baseline to four months and from baseline to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Intending to be available for a 24 month intervention

Exclusion Criteria:

* Unable to provide informed consent
* BMI < 18.5 kg/m2, >/=35 kg/m2
* Household member on study staff
* Past or planned (within the next 24 months) weight loss surgery (e.g. gastric bypass, lap band, or liposuction); current participation in a commercial weight loss program (e.g. Weight Watcher's, Jenny Craig); current or planned enrollment in another diet/physical activity/weight loss intervention study
* Regular use of systemic steroids, prescription weight loss drugs, and/or diabetes medications (oral or injected). "Regular use" is defined as "taking this medication most days of the week for the previous month"
* Current treatment for an eating disorder
* Cardiovascular event (heart attack, stroke, episode of heart failure, or revascularization procedure) within the last 6 months
* Current treatment for malignancy (other than non-melanoma skin cancer)
* Investigator discretion
* Currently pregnant or gave birth within the last 6 months, currently lactating or breastfeeding within the last 3 months, actively planning pregnancy within the next 24 months.
* Systolic BP at screening >/= 160 mmHg or diastolic BP >/= 100 mmHg. If BP exceeds this level, participants can return for re-screening after being evaluated and treated for hypertension.
* Weight loss of more than 15 lbs over the past three months
* Trying to gain weight.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 441 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa N. Laska, PhD, RD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - Anoka Ramsey Community College, Coon Rapids, Minnesota
  - Inver Hills Community College, Inver Grove Heights, Minnesota
  - Saint Paul College, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lytle LA, Laska MN, Linde JA, Moe SG, Nanney MS, Hannan PJ, Erickson DJ. Weight-Gain Reduction Among 2-Year College Students: The CHOICES RCT. Am J Prev Med. 2017 Feb;52(2):183-191. doi: 10.1016/j.amepre.2016.10.012. Epub 2016 Dec 6. PMID 27939237
- [Derived] Laska MN, Lytle LA, Nanney MS, Moe SG, Linde JA, Hannan PJ. Results of a 2-year randomized, controlled obesity prevention trial: Effects on diet, activity and sleep behaviors in an at-risk young adult population. Prev Med. 2016 Aug;89:230-236. doi: 10.1016/j.ypmed.2016.06.001. Epub 2016 Jun 7. PMID 27283096

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: 224 participants were randomized to the intervention condition
- Control Group: 217 participants were randomized to the control condition
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 224 | 217
Completed | 188 | 180
Not Completed | 36 | 37
Not completed — Pregnancy | 16 | 8
Not completed — Withdrawal by Subject | 15 | 9
Not completed — Lost to Follow-up | 5 | 20

BASELINE CHARACTERISTICS:
Population: The original study design was 4 arms (1 control & 3 intervention) that varied in the way the 4-month curriculum was delivered. Our formative work showed that students not being able to choose the course delivery method would limit interest in study participation. We changed the study design to 2 arms, which was approved by the EARLY trials DSMB.
Groups:
- Control Group: This control group arm consists of students who served as the comparison group.
- Intervention Group: This intervention arm is a combination of the face-to-face class students, hybrid class students and online class students
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 217 | 224 | 441
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 217 | 224 | 441
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 150 | 298
  Male | 69 | 74 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 33
  Not Hispanic or Latino | 201 | 207 | 408
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 14 | 13 | 27
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 40 | 28 | 68
  White | 149 | 171 | 320
  More than one race | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 217 | 224 | 441

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index (BMI)
Description: The primary aim of this study is to examine the effectiveness of a 24-month weight gain prevention intervention to positively affect body mass index (BMI) in 2-year college students. Our hypothesis is that students randomized to an intervention condition will experience a smaller increase in mean BMI post treatment as compared to students randomized to the control condition.
Time Frame: Baseline to 24 Months
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 179 | 187
kg/m2 | 26.2 (0.283) | 26.0 (0.280)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.707, Regression, Logistic — The analysis used hierarchical linear models having repeated measures of the outcome regressed on experimental condition, adjusted for baseline age, sex, race, and household education level as well as wave and college

2. Secondary Outcome: Prevalence of Overweight/Obese
Description: The prevalence of overweight/obese between intervention and control students
Time Frame: Baseline to 24 Months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 187 | 179
percentage of participants | 46.6 | 57.1
Statistical Analysis 1: Comparison: Control Group; Test type: Superiority or Other; p = 0.049, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change in BMI From Baseline to 4 Months
Description: Comparison of the effects of the intervention and control groups with regard to change in BMI from baseline to 4 months
Time Frame: Baseline to 4 Months
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 205 | 201
kg/m2 | 25.5 (0.273) | 25.6 (0.274)

4. Secondary Outcome: Change in Weight From Baseline to 4 Months
Description: Comparison of the effects of the intervention and control groups with regard to change in weight from baseline to 4 months
Time Frame: Baseline to 4 Months
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 205 | 201
Kg | 72.3 (0.834) | 72.7 (0.840)

5. Secondary Outcome: Change in BMI From Baseline to 12 Months
Description: Comparison of the effects of the intervention and control groups with regard to change in BMI from baseline to 12 months
Time Frame: Baseline to 12 Months
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 197 | 190
kg/m2 | 25.5 (0.274) | 25.7 (0.276)

6. Secondary Outcome: Change in Weight From Baseline to 12 Months
Description: Comparison of the effects of the intervention and control groups with regard to change in weight from baseline to 12 months
Time Frame: Baseline to 12 Months
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 197 | 190
Kg | 72.4 (0.839) | 73.1 (0.844)

ADVERSE EVENTS:
Time Frame: Baseline to 24 Months
Groups:
- Intervention Group: This intervention group is a combination of the face-to-face class students, hybrid class students and online class students.
- Control Group: This control group consists of students who served as the comparison group.
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 11/224 | 11/217
Other Adverse Events (participants affected / at risk) | 82/224 | 80/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=224) | Control Group (N=217)
CVD Events and Procedures (Cardiac disorders) | 1 (1) | 0 (0)
Fainting (General disorders) | 1 (1) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
Psychiatric (Psychiatric disorders) | 2 (2) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Motor Vehicle Accident (General disorders) | 1 (1) | 0 (0)
Other (General disorders) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=224) | Control Group (N=217)
CVD Events and Procedures (Cardiac disorders) | 0 (0) | 1 (1)
Fainting (General disorders) | 3 (3) | 9 (10)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 25 (25) | 21 (22)
Gall Bladder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Psychiatric (Psychiatric disorders) | 10 (11) | 16 (19)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Obstetric (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Motor Vehicle Accident (General disorders) | 10 (10) | 14 (15)
Other (General disorders) | 30 (30) | 15 (16)

LIMITATIONS AND CAVEATS:
Because of sample size constraints we combined overweight and obese participants into one category. Additional insights might be gleaned from examining intervention impact and transitions between three categories of weight status.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No